CLINICAL TRIAL: NCT02222077
Title: Diurnal Variation of Central Blood Pressure in Adolescents and Young Adults and Association With Indices of Asymptomatic Target-organ Damage
Brief Title: Central Blood Pressure in Adolescents and Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Professor of Medicine, University of Athens
Other Study IDs: Central BP-TOD
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Healthy; Hypertension
Keywords: Central blood pressure; Ambulatory blood pressure monitoring; Target-organ damage; Adolescents and young adults
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate in adolescents and young adults:

* the 24h diurnal variation of ambulatory central blood pressure
* the association of central compared to peripheral blood pressure with indices of asymptomatic target-organ damage

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults (age range 12-25 years)

Exclusion Criteria:

* Subjects with any acute or significant chronic disease, with evidence of secondary hypertension, or on regular drug treatment will be excluded

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy volunteers and subjects referred to the Hypertension Clinic for the assessment of elevated blood pressure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficients (r) between 24h ambulatory central blood pressure and indices of target-organ damage | Assessment of each individual will require up to 3 days
  Correlation coefficients (r) will be determined for the relationship between central blood pressure and indices of target-organ damage (left ventricular mass index, carotid intima-media thickness, pulse wave velocity). Also, these coefficients will be compared with z-statistic with the respective ones for the peripheral blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension Center, 3rd University Department of Medicine, Sotiria Hospital, Athens, Attica, Greece